CLINICAL TRIAL: NCT06304181
Title: Effect of Paracetamol and Mannitol Injection on Postoperative Analgesia in Patients With Thoracoscopic Lobectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY-2023-195
Record Dates: First submitted 2024-02-19; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Postoperative Analgesia
Keywords: Paracetamol and Mannitol Injection; postoperative analgesia; thoracic surgery
MeSH Terms: interventions — Acetaminophen; Mannitol; parecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paracetamol and Mannitol Injection group (Experimental): Paracetamol and Mannitol Injection 500mg was given intravenously 30 minutes before the end of the operation
  Interventions: Drug: Paracetamol and Mannitol Injection
- Parecoxib group (Active Comparator): 40mg of parecoxib was given intravenously 30min before the end of the operation
  Interventions: Drug: Parecoxib

INTERVENTIONS:
Drug: Paracetamol and Mannitol Injection — Paracetamol and Mannitol Injection 500mg
  Other Names: Acetaminophen Mannitol Injection
  Arms: Paracetamol and Mannitol Injection group
Drug: Parecoxib — 40mg of parecoxib
  Arms: Parecoxib group

SUMMARY:
This study thoroughly evaluates the efficacy of acetaminophen mannitol injection for postoperative analgesia in patients undergoing thoracoscopic lobectomy, by comparing it with a control group.

ELIGIBILITY:
Inclusion Criteria:

1. Obtain informed consent；
2. Patients scheduled for partial lobectomy under thoracoscopy with general anesthesia；
3. Classified as American Society of Anesthesiologists (ASA) physical status I~II；
4. Age over 18 years；
5. Patients voluntarily participate and sign the informed consent form

Exclusion Criteria:

1. Systolic blood pressure ≥180 mm Hg or <90 mm Hg, diastolic blood pressure ≥110 mm Hg or <60 mmHg
2. heart rate <50 beats/min；
3. Patients with severe liver or kidney dysfunction (severe liver dysfunction: ALT, conjugated bilirubin, AST, ALP, total bilirubin any one >2 times the upper limit of normal
4. severe kidney dysfunction: creatinine clearance <60 ml/min)；
5. Patients with diabetes and complications (diabetic ketoacidosis, hyperosmolar coma, various infections, major vascular changes, diabetic nephropathy, retinopathy, diabetic cardiomyopathy, diabetic neuropathy, diabetic foot, etc.)；
6. Patients with severe pulmonary impairment, such as asthma or chronic obstructive pulmonary disease；
7. History of psychiatric illness or long-term use of psychiatric drugs, chronic pain medication, or history of alcohol abuse；
8. Neuromuscular diseases；
9. Tendency towards malignant hyperthermia；
10. Allergy to the study drug or other contraindications；
11. Participation in another drug clinical trial within the past 30 days；
12. Any cerebrovascular accidents such as stroke, transient ischemic attack (TIA) in the last 3 months；
13. Unstable angina, myocardial infarction in the last 3 months；
14. Undergone another surgery within the last 3 months；
15. Coagulopathy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
NRS scores | after extubation 10 (±5) minutes, before leaving the resuscitation room, 6 hours, 12 hours, 24 hours after surgery
  NRS scores at rest and during movement (coughing) after extubation 10 (±5) minutes, before leaving the resuscitation room, 6 hours, 12 hours, 24 hours after surgery
RASS score | after extubation 10 (±5) minutes and 24 hours after surgery
  RASS score after extubation 10 (±5) minutes and 24 hours after surgery

SECONDARY OUTCOMES:
Time of first use of remedial analgesics or analgesic pump | From the end of surgery until the date of first use of remedial analgesics or analgesic pumps,assessed up to 3 days
  Time of first use of remedial analgesics or analgesic pump after surgery,assessed up to 3 days
Total analgesic pump drug use | From the end of surgery until removal of the analgesic pump,assessed up to 3 days
  The total drug use of analgesic pump was recorded during follow-up
Postoperative liver enzyme level | Time 1 (Within 5 minutes of the surgery), Time 2 (1 day post-surgery), Time 3 (2 days post-surgery)
  Measurement of level of liver enzymes in the blood in Time 1 (Within 5 minutes of the surgery), Time 2 (1 day post-surgery), Time 3 (2 days post-surgery)
Postoperative bilirubin level | Time 1 (Within 5 minutes of the surgery), Time 2 (1 day post-surgery), Time 3 (2 days post-surgery)
  Measurement of level of bilirubin in the blood in Time 1 (Within 5 minutes of the surgery), Time 2 (1 day post-surgery), Time 3 (2 days post-surgery)
Postoperative creatinine level | Time 1 (Within 5 minutes of the surgery), Time 2 (1 day post-surgery), Time 3 (2 days post-surgery)
  Measurement of level of creatinine in the blood in Time 1 (Within 5 minutes of the surgery), Time 2 (1 day post-surgery), Time 3 (2 days post-surgery)
Postoperative cortisol level | Time 1 (Within 5 minutes of the surgery), Time 2 (1 day post-surgery), Time 3 (2 days post-surgery)
  Measurement of level of ccortisol in the blood in Time 1 (Within 5 minutes of the surgery), Time 2 (1 day post-surgery), Time 3 (2 days post-surgery)
Postoperative IL-6 level | Time 1 (Within 5 minutes of the surgery), Time 2 (1 day post-surgery), Time 3 (2 days post-surgery)
  Measurement of level of IL-6 in the blood in Time 1 (Within 5 minutes of the surgery), Time 2 (1 day post-surgery), Time 3 (2 days post-surgery)
Postoperative IL-8 level | Time 1 (Within 5 minutes of the surgery), Time 2 (1 day post-surgery), Time 3 (2 days post-surgery)
  Measurement of level of IL-8 in the blood in Time 1 (Within 5 minutes of the surgery), Time 2 (1 day post-surgery), Time 3 (2 days post-surgery)

IPD SHARING:
Plan to Share IPD: No